CLINICAL TRIAL: NCT00839397
Title: BRL29060A in Posttraumatic Stress Disorder
Brief Title: BRL29060A (Paroxetine Hydrochloride Hydrate) in Posttraumatic Stress Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 29060/799
Record Dates: First submitted 2009-01-29; First posted 2009-02-09 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2014-03

CONDITIONS: Post-Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Paroxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paroxetine (Other): A 52-week, non-comparative, uncontrolled study (However, the baseline phase is single blind)
  Interventions: Drug: Paroxetine

INTERVENTIONS:
Drug: Paroxetine — Subjects will take the treatment phase medication once daily after an evening meal. All subjects will be maintained at Dose Level II (20 mg/day) for the first 2 weeks. If a sufficient clinical response ("1. Very much improved" or "2. Much improved" based on the CGI Global Improvement) is achieved, the subject will continue on the same dose level. When the clinical response is not sufficient but the investigational product is well tolerated, the dose will be increased to Dose Level III (30 mg/day) and then to Dose Level IV (40 mg/day) at intervals of at least 2 weeks until a sufficient response is reached. Once a sufficient response is obtained, the treatment will be continued at that dose. The treatment phase will last for a total of 52 weeks. In those patients receiving Dose Level III or IV, dosage reductions to the next lowest level (Dose Level II or III) consequent to an adverse event are permitted.
  Dosage adjustment will be made at the discretion of the PI or Sub-PI

SUMMARY:
This was a 52-week, non-comparative, uncontrolled study of paroxetine in Japanese PTSD patients to obtain clinical experience regarding efficacy and safety. In this study, subjects received paroxetine 20mg-40mg once daily after an evening meal.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a primary diagnosis of PTSD according to DSM-IV criteria (Posttraumatic Stress Disorder: 309.81). In order to diagnose PTSD, the Clinician-Administered PTSD Scale-DX Current and Lifetime Diagnostic Version (CAPS-DX) will be used.
* Disease to Be Treated:
* Duration of illness of at least 3 months at Week -1.
* Score >= 50 on Criteria B, C and D of CAPS-SX.
* Age: >=18 - <65 years (at the time of acquisition of informed consent)
* Sex: No restriction
* Hospitalization Status: No restriction
* Informed consent: Gives his/her informed consent. In case of a subject who is under the age of 20, his/her parent/guardian must also give his/her written informed consent.

Exclusion Criteria:

Exclusion Criteria at Week -1

* Patients diagnosed with Axis I disorders (excluding PTSD) such as major depression, dysthymia, simple phobia, OCD, or panic disorder as a primary diagnosis according to DSM-IV criteria within 24 weeks prior to Week -1. However, patients with depressive disorders are allowed to enroll in the study, if PTSD was present before the depressive disorders appeared and PTSD is the predominant disorder.
* Patients presenting a current major depressive episode that preceded the diagnosis of PTSD. However, patients with depressive disorders are allowed to enroll in the study, if PTSD was present before the depressive disorders appeared and PTSD is the predominant disorder.
* Patients receiving disability payments because of PTSD or any other psychiatric disorder.
* Patients currently engaged in compensation litigation whereby personal gain would be achieved from prolonged symptoms of PTSD or any other psychiatric disorders.
* Patients taking St. Johns Wort.
* Patients who meet DSM-IV criteria for substance abuse (alcohol or drugs) or substance dependence within 24 weeks prior to Week -1.
* Patients who have attempted suicide within 24 weeks prior to Week -1 or who pose, in the investigator's judgement using the M.I.N.I. "C. Suicidality", a high suicidal risk.
* Women who are pregnant or lactating, who may be pregnant, or who plan for pregnancy during the study.
* Patients who have taken MAO inhibitors within 1 week prior to Week -1 (or within 2 weeks prior to Week 0).
* Patients who have had electroconvulsive therapy (ECT) within 12 weeks prior to Week -1.
* Patients who have been treated with another investigational drug within 12 weeks prior to Week -1.
* Patients with a history or complication of manic psychosis.
* Patients with a history or complication of convulsive disorder (epilepsy, etc.).
* Patients with a complication of glaucoma.
* Patients with a known tendency for bleeding or those with predisposing conditions.
* Patients with a history of hypersensitivity to paroxetine.
* Patients with any serious organic disorder in the brain.
* Patients with any serious physical symptom such as cardiac, hepatic, renal or hematopoietic dysfunction.
* Patients with a history or complication of cancer or malignant tumor.
* Others whom the investigator or sub-investigator considers ineligible for the study.

Exclusion Criterion at Week 0

* Patients whose placebo run-in medication compliance is less than 80%.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2002-05; Primary Completion 2004-11 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Clinician-Administered Posttraumatic Stress Disorder Scale One Week Symptom Status Version (CAPS-SX) total score | 52 weeks

SECONDARY OUTCOMES:
Proportion of responders based on the CGI Global Improvement | 52 weeks
Change from baseline in the CAPS-SX re-experiencing cluster score | 52 weeks
Change from baseline in the CAPS-SX avoidance/numbing cluster score | 52 weeks
Change from baseline in the CAPS-SX hyperarousal cluster score | 52 weeks
Change from baseline in the CGI Severity of Illness score | 52 weeks
Adverse events (AEs), abnormal findings in each examination/test, and their details: Laboratory tests (hematology, clinical chemistry, electrolytes, urinalysis), Blood pressure, pulse rate, body weight | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Background] Kim Y, Asukai N, Konishi T, Kato H, Hirotsune H, Maeda M, Inoue H, Narita H, Iwasaki M. Clinical evaluation of paroxetine in post-traumatic stress disorder (PTSD): 52-week, non-comparative open-label study for clinical use experience. Psychiatry Clin Neurosci. 2008 Dec;62(6):646-52. doi: 10.1111/j.1440-1819.2008.01862.x. PMID 19068000